CLINICAL TRIAL: NCT03059979
Title: Hit Hard and Early. The Effect of High Dose Methylprednisolone on Nailfold Capillary Changes and Biomarkers in Early SSc: a 12-week Randomised Explorative Double-blind Placebo-controlled Trial.
Brief Title: The Effect of High Dose Methylprednisolone on Nailfold in Early Systemic Sclerosis ( SSc )
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HHaE
Record Dates: First submitted 2017-01-25; First posted 2017-02-23 (Actual); Last update posted 2019-11-29 (Actual); Status verified 2019-09

CONDITIONS: Systemic Sclerosis; Raynaud Phenomena
MeSH Terms: conditions — Scleroderma, Systemic | interventions — Methylprednisolone; Methylprednisolone Hemisuccinate; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Methylprednisolone 1000 mg (Active Comparator): the methylprednisolone is dissolved in 100 cc of sodium chloride (NaCl 0.9%) by intravenous infusion in 30 minutes on three consecutive days
  Interventions: Drug: Methylprednisolone
- sodium chloride (Placebo Comparator): The placebo intervention with physiologic salt solution is identical in appearance
  Interventions: Other: sodium chloride

INTERVENTIONS:
Drug: Methylprednisolone — methylprednisolone 1000 mg dissolved in 100 cc of NaCl 0.9%, by intravenous infusion in 30 minutes on three consecutive days Three-day treatment courses are given at week 0, week 4 and week 8.
  Other Names: Solu-Medrol
  Arms: Methylprednisolone 1000 mg
Other: sodium chloride — 100 cc of NaCl 0,9% , administered by intravenous infusion in 30 minutes on three consecutive days Three-day treatment courses are given at week 0, week 4 and week 8.
  Other Names: NaCl 0,9%
  Arms: sodium chloride

SUMMARY:
This is a 12 week double-blind randomized placebo controlled trial in which 30 patients with very early SSc, fulfilling the Very Early Diagnosis Of Systemic Sclerosis (VEDOSS) criteria (9) will be randomized in a 2:1 fashion to receive intravenous methylprednisolone or placebo. Three-day treatment courses are given at week 0, week 4 and week 8. The final assessment is at week 12, and patients will be followed up to one year after baseline

DETAILED DESCRIPTION:
Systemic sclerosis is a disease with a high burden caused by morbidity and increased mortality. To date a cure for SSc is not available. In this trial, patients are treated very early in the disease which could change the long term outcome of SSc in these patients.

In daily practice, patients so early in the disease course are not treated although they might be at risk for early escalation and internal organ involvement, reducing their prognosis. A trial to investigate the efficacy of a relative save, inexpensive and easy accessible treatment will provide us with the opportunity to change the disease course and reducing the disease burden of a portion of the SSc patients

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Age over 18 years
* Fulfilling VEDOSS criteria (9):

  * Raynauds' Phenomenon and
  * Positive for disease specific auto antibodies (anti-centromere or anti-topoisomerase antibodies) and
  * typical nail fold capillaroscopic findings
* Puffy fingers < 3 years
* Modified Rodnan skin score = 0

Exclusion Criteria:

* Presence of acroosclerosis, acrosteolysis and digital ulcers
* Presence of anti-RNA polymerase III auto antibodies

Previous systemic treatment for SSc, namely:

* methotrexate,
* prednisone (> 14 days in previous 6 months),
* mofetil mycophenolate
* cyclophosphamide.

Clinically significant internal organ involvement:

* diffusion capacity of lung for carbon monoxide (DLCO) < 80% predicted,
* vital capacity (VC) < 70% predicted
* renal dysfunction with glomerular filtration rate (GFR) < 60 ml/min
* diastolic dysfunction > grade 1 on echocardiography
* pulmonary hypertension
* weight loss >10% in the last 6 months with unknown cause

Contra-indications for methylprednisolone, such as:

* pregnancy, lactation
* psychotic or depressive disorder
* ulcus duodeni or ventriculi
* untreated hypertension (> 160-90 mmHg)
* acute infections

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-01; Primary Completion 2021-07-01 (Estimated); Study Completion 2021-07-01 (Estimated)

PRIMARY OUTCOMES:
the change in capillary density from baseline | 12 weeks
  presence of enlarged and giant capillaries, hemorrhages, loss of capillaries, disorganization of the micro vascular array, and capillary ramifications.

SECONDARY OUTCOMES:
change in selected biomarkers: the interferon signature in peripheral blood from baseline | 1 year
  Plasma biomarkers consist soluble inflammatory mediators platelet factor 4, interleukin-1β, interleukin-6, tumor necrosis factor-α, endothelin-1, intercellular adhesion molecule-1 and vascular endothelial growth factor
change in nail fold capillary changes other than capillary density and giant capillaries from baseline | 1 year
  changes in nail fold capillary pattern (early, active, late, normal
change in modified Rodnan skin score (mRSS) from baseline | 1 year
presence of puffy fingers from baseline | 1 year
presence of synovitis from baseline | 1 year
presence of tendon friction rubs from baseline | 1 year
fulfilling EULAR/ACR ( American College of Rheumatology )classification from baseline criteria for SSc from baseline | 1 year
pulmonary function tests from baseline | 1 year
presence of interstitial lung disease from baseline | 1 year
suspicion of pulmonary hypertension from baseline | 1 year
Change in physical function from baseline | 1 year
general health score from baseline | 1 year
Change in 36-Item Short Form Survey (SF-36) total score from baseline | 1 year
Change in Scleroderma Health Assessment Questionnaire (SHAQ)total score from baseline | 1 year
Change in EQ-5D is a standardised instrument for use as a measure of health outcome. (EQ5D) total score from baseline | 1 year
Change in gastrointestinal tract ( GIT ) total score from baseline | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Madelon Vonk, Dr., Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboudumc, Rheumatology department, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Geyer M, Muller-Ladner U. The pathogenesis of systemic sclerosis revisited. Clin Rev Allergy Immunol. 2011 Apr;40(2):92-103. doi: 10.1007/s12016-009-8193-3. PMID 20087791
- [Background] van Bon L, Affandi AJ, Broen J, Christmann RB, Marijnissen RJ, Stawski L, Farina GA, Stifano G, Mathes AL, Cossu M, York M, Collins C, Wenink M, Huijbens R, Hesselstrand R, Saxne T, DiMarzio M, Wuttge D, Agarwal SK, Reveille JD, Assassi S, Mayes M, Deng Y, Drenth JP, de Graaf J, den Heijer M, Kallenberg CG, Bijl M, Loof A, van den Berg WB, Joosten LA, Smith V, de Keyser F, Scorza R, Lunardi C, van Riel PL, Vonk M, van Heerde W, Meller S, Homey B, Beretta L, Roest M, Trojanowska M, Lafyatis R, Radstake TR. Proteome-wide analysis and CXCL4 as a biomarker in systemic sclerosis. N Engl J Med. 2014 Jan 30;370(5):433-43. doi: 10.1056/NEJMoa1114576. Epub 2013 Dec 18. PMID 24350901
- [Background] Radstake TR, Gorlova O, Rueda B, Martin JE, Alizadeh BZ, Palomino-Morales R, Coenen MJ, Vonk MC, Voskuyl AE, Schuerwegh AJ, Broen JC, van Riel PL, van 't Slot R, Italiaander A, Ophoff RA, Riemekasten G, Hunzelmann N, Simeon CP, Ortego-Centeno N, Gonzalez-Gay MA, Gonzalez-Escribano MF; Spanish Scleroderma Group; Airo P, van Laar J, Herrick A, Worthington J, Hesselstrand R, Smith V, de Keyser F, Houssiau F, Chee MM, Madhok R, Shiels P, Westhovens R, Kreuter A, Kiener H, de Baere E, Witte T, Padykov L, Klareskog L, Beretta L, Scorza R, Lie BA, Hoffmann-Vold AM, Carreira P, Varga J, Hinchcliff M, Gregersen PK, Lee AT, Ying J, Han Y, Weng SF, Amos CI, Wigley FM, Hummers L, Nelson JL, Agarwal SK, Assassi S, Gourh P, Tan FK, Koeleman BP, Arnett FC, Martin J, Mayes MD. Genome-wide association study of systemic sclerosis identifies CD247 as a new susceptibility locus. Nat Genet. 2010 May;42(5):426-9. doi: 10.1038/ng.565. Epub 2010 Apr 11. PMID 20383147
- [Background] Greenblatt MB, Aliprantis AO. The immune pathogenesis of scleroderma: context is everything. Curr Rheumatol Rep. 2013 Jan;15(1):297. doi: 10.1007/s11926-012-0297-8. PMID 23288576
- [Background] Tyndall AJ, Bannert B, Vonk M, Airo P, Cozzi F, Carreira PE, Bancel DF, Allanore Y, Muller-Ladner U, Distler O, Iannone F, Pellerito R, Pileckyte M, Miniati I, Ananieva L, Gurman AB, Damjanov N, Mueller A, Valentini G, Riemekasten G, Tikly M, Hummers L, Henriques MJ, Caramaschi P, Scheja A, Rozman B, Ton E, Kumanovics G, Coleiro B, Feierl E, Szucs G, Von Muhlen CA, Riccieri V, Novak S, Chizzolini C, Kotulska A, Denton C, Coelho PC, Kotter I, Simsek I, de la Pena Lefebvre PG, Hachulla E, Seibold JR, Rednic S, Stork J, Morovic-Vergles J, Walker UA. Causes and risk factors for death in systemic sclerosis: a study from the EULAR Scleroderma Trials and Research (EUSTAR) database. Ann Rheum Dis. 2010 Oct;69(10):1809-15. doi: 10.1136/ard.2009.114264. Epub 2010 Jun 15. PMID 20551155
- [Background] Kowal-Bielecka O, Landewe R, Avouac J, Chwiesko S, Miniati I, Czirjak L, Clements P, Denton C, Farge D, Fligelstone K, Foldvari I, Furst DE, Muller-Ladner U, Seibold J, Silver RM, Takehara K, Toth BG, Tyndall A, Valentini G, van den Hoogen F, Wigley F, Zulian F, Matucci-Cerinic M; EUSTAR Co-Authors. EULAR recommendations for the treatment of systemic sclerosis: a report from the EULAR Scleroderma Trials and Research group (EUSTAR). Ann Rheum Dis. 2009 May;68(5):620-8. doi: 10.1136/ard.2008.096677. Epub 2009 Jan 15. PMID 19147617
- [Background] van Laar JM, Farge D, Sont JK, Naraghi K, Marjanovic Z, Larghero J, Schuerwegh AJ, Marijt EW, Vonk MC, Schattenberg AV, Matucci-Cerinic M, Voskuyl AE, van de Loosdrecht AA, Daikeler T, Kotter I, Schmalzing M, Martin T, Lioure B, Weiner SM, Kreuter A, Deligny C, Durand JM, Emery P, Machold KP, Sarrot-Reynauld F, Warnatz K, Adoue DF, Constans J, Tony HP, Del Papa N, Fassas A, Himsel A, Launay D, Lo Monaco A, Philippe P, Quere I, Rich E, Westhovens R, Griffiths B, Saccardi R, van den Hoogen FH, Fibbe WE, Socie G, Gratwohl A, Tyndall A; EBMT/EULAR Scleroderma Study Group. Autologous hematopoietic stem cell transplantation vs intravenous pulse cyclophosphamide in diffuse cutaneous systemic sclerosis: a randomized clinical trial. JAMA. 2014 Jun 25;311(24):2490-8. doi: 10.1001/jama.2014.6368. PMID 25058083
- [Background] Czirjak L, Matucci-Cerinic M. Beyond Raynaud's phenomenon hides very early systemic sclerosis: the assessment of organ involvement is always mandatory. Rheumatology (Oxford). 2011 Feb;50(2):250-1. doi: 10.1093/rheumatology/keq374. Epub 2010 Nov 28. No abstract available. PMID 21115465
- [Background] Minier T, Guiducci S, Bellando-Randone S, Bruni C, Lepri G, Czirjak L, Distler O, Walker UA, Fransen J, Allanore Y, Denton C, Cutolo M, Tyndall A, Muller-Ladner U, Matucci-Cerinic M; EUSTAR co-workers; EUSTAR co-workers. Preliminary analysis of the very early diagnosis of systemic sclerosis (VEDOSS) EUSTAR multicentre study: evidence for puffy fingers as a pivotal sign for suspicion of systemic sclerosis. Ann Rheum Dis. 2014 Dec;73(12):2087-93. doi: 10.1136/annrheumdis-2013-203716. Epub 2013 Aug 12. PMID 23940211
- [Background] Hahn BH, Kantor OS, Osterland CK. Azathioprine plus prednisone compared with prednisone alone in the treatment of systemic lupus erythematosus. Report of a prospective controlled trial in 24 patients. Ann Intern Med. 1975 Nov;83(5):597-605. doi: 10.7326/0003-4819-83-5-597. PMID 1106277
- [Background] Marie I, Mouthon L. Therapy of polymyositis and dermatomyositis. Autoimmun Rev. 2011 Nov;11(1):6-13. doi: 10.1016/j.autrev.2011.06.007. Epub 2011 Jun 28. PMID 21740984
- [Background] Rhen T, Cidlowski JA. Antiinflammatory action of glucocorticoids--new mechanisms for old drugs. N Engl J Med. 2005 Oct 20;353(16):1711-23. doi: 10.1056/NEJMra050541. No abstract available. PMID 16236742
- [Background] Iudici M, van der Goes MC, Valentini G, Bijlsma JW. Glucocorticoids in systemic sclerosis: weighing the benefits and risks - a systematic review. Clin Exp Rheumatol. 2013 Mar-Apr;31(2 Suppl 76):157-65. Epub 2013 Jul 23. PMID 23910618
- [Background] Matucci-Cerinic M, Bellando-Randone S, Lepri G, Bruni C, Guiducci S. Very early versus early disease: the evolving definition of the 'many faces' of systemic sclerosis. Ann Rheum Dis. 2013 Mar;72(3):319-21. doi: 10.1136/annrheumdis-2012-202295. Epub 2012 Nov 23. No abstract available. PMID 23178210
- [Background] Auphan N, DiDonato JA, Rosette C, Helmberg A, Karin M. Immunosuppression by glucocorticoids: inhibition of NF-kappa B activity through induction of I kappa B synthesis. Science. 1995 Oct 13;270(5234):286-90. doi: 10.1126/science.270.5234.286. PMID 7569976
- [Background] Davies CA, Jeziorska M, Freemont AJ, Herrick AL. The differential expression of VEGF, VEGFR-2, and GLUT-1 proteins in disease subtypes of systemic sclerosis. Hum Pathol. 2006 Feb;37(2):190-7. doi: 10.1016/j.humpath.2005.10.007. Epub 2005 Dec 15. PMID 16426919
- [Background] Stratton RJ, Coghlan JG, Pearson JD, Burns A, Sweny P, Abraham DJ, Black CM. Different patterns of endothelial cell activation in renal and pulmonary vascular disease in scleroderma. QJM. 1998 Aug;91(8):561-6. doi: 10.1093/qjmed/91.8.561. PMID 9893759
- [Background] Greenberg SA, Higgs BW, Morehouse C, Walsh RJ, Kong SW, Brohawn P, Zhu W, Amato A, Salajegheh M, White B, Kiener PA, Jallal B, Yao Y. Relationship between disease activity and type 1 interferon- and other cytokine-inducible gene expression in blood in dermatomyositis and polymyositis. Genes Immun. 2012 Apr;13(3):207-13. doi: 10.1038/gene.2011.61. Epub 2011 Sep 1. PMID 21881594
- [Background] Higgs BW, Liu Z, White B, Zhu W, White WI, Morehouse C, Brohawn P, Kiener PA, Richman L, Fiorentino D, Greenberg SA, Jallal B, Yao Y. Patients with systemic lupus erythematosus, myositis, rheumatoid arthritis and scleroderma share activation of a common type I interferon pathway. Ann Rheum Dis. 2011 Nov;70(11):2029-36. doi: 10.1136/ard.2011.150326. Epub 2011 Jul 28. PMID 21803750
- [Background] Miniati I, Guiducci S, Conforti ML, Rogai V, Fiori G, Cinelli M, Saccardi R, Guidi S, Bosi A, Tyndall A, Matucci-Cerinic M. Autologous stem cell transplantation improves microcirculation in systemic sclerosis. Ann Rheum Dis. 2009 Jan;68(1):94-8. doi: 10.1136/ard.2007.082495. Epub 2008 Feb 28. PMID 18308744
- [Background] Hunzelmann N, Moinzadeh P, Genth E, Krieg T, Lehmacher W, Melchers I, Meurer M, Muller-Ladner U, Olski TM, Pfeiffer C, Riemekasten G, Schulze-Lohoff E, Sunderkoetter C, Weber M; German Network for Systemic Scleroderma Centers. High frequency of corticosteroid and immunosuppressive therapy in patients with systemic sclerosis despite limited evidence for efficacy. Arthritis Res Ther. 2009;11(2):R30. doi: 10.1186/ar2634. Epub 2009 Mar 4. PMID 19261182
- [Background] Smith V, Decuman S, Sulli A, Bonroy C, Piettte Y, Deschepper E, de Keyser F, Cutolo M. Do worsening scleroderma capillaroscopic patterns predict future severe organ involvement? a pilot study. Ann Rheum Dis. 2012 Oct;71(10):1636-9. doi: 10.1136/annrheumdis-2011-200780. Epub 2012 Mar 8. PMID 22402146
- [Background] Valentini G, Marcoccia A, Cuomo G, Vettori S, Iudici M, Bondanini F, Santoriello C, Ciani A, Cozzolino D, De Matteis GM, Cappabianca S, Vitelli F, Spano A. Early systemic sclerosis: analysis of the disease course in patients with marker autoantibody and/or capillaroscopic positivity. Arthritis Care Res (Hoboken). 2014 Oct;66(10):1520-7. doi: 10.1002/acr.22304. PMID 24515450
- [Background] van den Hoogen F, Khanna D, Fransen J, Johnson SR, Baron M, Tyndall A, Matucci-Cerinic M, Naden RP, Medsger TA Jr, Carreira PE, Riemekasten G, Clements PJ, Denton CP, Distler O, Allanore Y, Furst DE, Gabrielli A, Mayes MD, van Laar JM, Seibold JR, Czirjak L, Steen VD, Inanc M, Kowal-Bielecka O, Muller-Ladner U, Valentini G, Veale DJ, Vonk MC, Walker UA, Chung L, Collier DH, Ellen Csuka M, Fessler BJ, Guiducci S, Herrick A, Hsu VM, Jimenez S, Kahaleh B, Merkel PA, Sierakowski S, Silver RM, Simms RW, Varga J, Pope JE. 2013 classification criteria for systemic sclerosis: an American college of rheumatology/European league against rheumatism collaborative initiative. Ann Rheum Dis. 2013 Nov;72(11):1747-55. doi: 10.1136/annrheumdis-2013-204424. PMID 24092682
- [Background] Tan FK, Zhou X, Mayes MD, Gourh P, Guo X, Marcum C, Jin L, Arnett FC Jr. Signatures of differentially regulated interferon gene expression and vasculotrophism in the peripheral blood cells of systemic sclerosis patients. Rheumatology (Oxford). 2006 Jun;45(6):694-702. doi: 10.1093/rheumatology/kei244. Epub 2006 Jan 17. PMID 16418202
- [Background] Cutolo M, Sulli A, Pizzorni C, Accardo S. Nailfold videocapillaroscopy assessment of microvascular damage in systemic sclerosis. J Rheumatol. 2000 Jan;27(1):155-60. PMID 10648032
- [Derived] Kersten BE, Lemmers JMJ, Vanhaecke A, Velauthapillai A, van den Hombergh WMT, van den Hoogen FHJ, van den Ende CHM, Smith V, Vonk MC. Efficacy of methylprednisolone in very early systemic sclerosis: results of the 'Hit Hard and Early' randomized controlled trial. Rheumatology (Oxford). 2025 Mar 1;64(3):1261-1269. doi: 10.1093/rheumatology/keae156. PMID 38552324
- [Derived] van den Hombergh WMT, Kersten BE, Knaapen-Hans HKA, Thurlings RM, van der Kraan PM, van den Hoogen FHJ, Fransen J, Vonk MC. Hit hard and early: analysing the effects of high-dose methylprednisolone on nailfold capillary changes and biomarkers in very early systemic sclerosis: study protocol for a 12-week randomised controlled trial. Trials. 2018 Aug 22;19(1):449. doi: 10.1186/s13063-018-2798-x. PMID 30134971